CLINICAL TRIAL: NCT01600326
Title: A Prospective Comparison of Ultrasound-Guided Percutaneous Platelet-Rich Plasma Injection Versus Tenotomy for Treatment of Gluteus Minimus and Medius Tendinosis
Brief Title: A Prospective Comparison of Ultrasound-Guided Percutaneous Platelet-Rich Plasma Injection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jon Jacobson, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00039445
Record Dates: First submitted 2012-05-01; First posted 2012-05-17 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-02

CONDITIONS: Tendinosis; Tendinitis
MeSH Terms: conditions — Tendinopathy | interventions — Tenotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tenotomy Group (Active Comparator): Subject enrolled in this arm will receive treatment for tendinitis and pain evaluation of pain pre and post treatment.
  Interventions: Procedure: Tenotomy (no injection)
- Plasma Injection Group (Active Comparator): Treatment is Ultrasound guided platelet rich plasma injection.
  Interventions: Drug: Ultrasound guided platelet rich plasma injection

INTERVENTIONS:
Procedure: Tenotomy (no injection) — Subjects randomized to this group will fill out a pre-treatment pain survey and have a blood draw They will be be contacted by the investigator by telephone or email on day 7 and day 14 to complete another pain survey. Subjects must avoid non steroidal anti-inflammatory medications for 2 weeks before the study. Two weeks after enrollment subjects see their referring physician to begin physical therapy.
  Arms: Tenotomy Group
Drug: Ultrasound guided platelet rich plasma injection — Subjects will fill out a pre-treatment pain survey, then will undergo ultrasound and have blood drawn from their arm.
  The blood sample will be separated into blood cells and plasma. The plasma portion of the blood (liquid minus the cells) will be injected into the tendon under sterile conditions. Ultrasound will help guide the injection. This is called "Ultrasound guided platelet rich plasma injection."
  Subjects will be be contacted by the investigator by telephone or email on day 7 and day 14 to complete another pain survey. Subjects must avoid non steroidal anti inflammatory medications for 2 weeks before the study and 2 weeks after the study.
  Subjects will see their referring physician two weeks after treatment to begin physical therapy.
  Arms: Plasma Injection Group

SUMMARY:
The purpose of this study is to determine the effectiveness of various treatment soft tendinosis also known as tendinitis.

DETAILED DESCRIPTION:
Currently there are three treatments that are considered standard of care; rest, tenotomy and tenotomy with injections of platelet-rich plasma (PRP). Tenotomy is performed by passing a needle through the abnormal tendon repeatedly until the needle has passed through all areas of the abnormal tendon with softening of the tendon. Tenotomy with PRP injections is performed in the same manner but includes an injection of platelet-rich plasma (PRP) into the tendon. This study will evaluate the effectiveness of tenotomy versus PRP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with a diagnosis of tendinosis of the hip.
* Adult subjects who have been referred to Dr. Jacobson for the treatment of tendinosis by tenotomy.

Exclusion Criteria:

* pregnancy
* risk of bleeding due to anticoagulant medication
* presence of malignancy
* steroid injection less than 3 months before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Jacobson, MD, Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Plasma Injection Group: Treatment is Ultrasound guided platelet rich plasma injection.
  Ultrasound guided platelet rich plasma injection: Subjects will fill out a pre-treatment pain survey, then will undergo ultrasound and have blood drawn from their arm.
  The blood sample will be separated into blood cells and plasma. The plasma portion of the blood (liquid minus the cells) will be injected into the tendon under sterile conditions. Ultrasound will help guide the injection. This is called "Ultrasound guided platelet rich plasma injection."
  Subjects will be be contacted by the investigator by telephone or email on day 7 and day 14 to complete another pain survey. Subjects must avoid non steroidal anti inflammatory medications for 2 weeks before the study and 2 weeks after the study.
  Subjects will see their referring physician two weeks after treatment to begin physical therapy.
Period: Overall Study
Arm/Group | Tenotomy Group | Plasma Injection Group
Started | 15 | 15
Primary Outcome Measure Data Collection | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenotomy Group | Plasma Injection Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Full Range); unit: years] | 60 [31 to 81] | 53 [24 to 72] | 57 [24 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
50 Point Pain and Interfence with Activity scale [Mean (Full Range); unit: units on a scale] — 50 Point Pain and Interfence with Activity scale with 0 as no pain or interference
  units on a scale | 32.4 [8 to 49] | 31.4 [11 to 41] | 31.9 [8 to 49]

OUTCOME MEASURES:

1. Primary Outcome: Pain Level and Interference With Activity
Description: Patient symptoms are measured on a 50 point scale where 0 is no pain or interference with activities and 50 is highest pain and interference.
  A verbal evaluation and assessment of subject's pain and symptoms will be completed prior to treatment. After receiving medication a second evaluation will be taken to determine how well the medication has relieved and controlled the subject's pain and inflammation associated with tendinitis.
  Subjects will be specifically asked to rate the level of pain and how the pain is affecting common activities of daily living. The outcomes will be assessed at 2 follow up periods, 1 and approximately 2 weeks after treatment (but no more than 23 days).
Time Frame: Up to 23 days
Population: One data point is missing for time point one for Plasma Injection Group, as noted below.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Tenotomy Group | Plasma Injection Group
Number analyzed (Participants) | 15 | 15
units on a scale
  1 week after treatment: number analyzed (Participants) | 15 | 14
  1 week after treatment | 16.8 [0 to 34] | 25.5 [9 to 41]
  2 wks post treatment ( no more than 23 days) | 15.2 [0 to 34] | 19.4 [4 to 42]
Statistical Analysis 1: Comparison: Tenotomy Group vs Plasma Injection Group; Test type: Other — Pair-wise comparison at Time point 1 compared to baseline; p < 0.0001, Tukey — One way repeated measure analysis of variance for outcome of total pain score over time adjusted for treatment with post hoc Tukey correction to adjust for multiple comparison; See comments on P value
Statistical Analysis 2: Comparison: Tenotomy Group vs Plasma Injection Group; One way repeated measure analysis of variance for outcome of total pain score over time adjusted for treatment with post hoc Tukey correction to adjust for multiple comparison; Test type: Superiority; p < 0.0001, Tukey — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants Showing Symptomatic Improvement as Assessed in Patient Chart
Description: Information from patient charts were retrospectively reviewed to determine if symptoms were reported as improved, worse, or no change over a time period (range 15 to 555 days post treatment).
Time Frame: 15 to 555 days post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Tenotomy Group | Plasma Injection Group
Number analyzed (Participants) | 14 | 14
Participants | 10 | 11
Statistical Analysis 1: Comparison: Tenotomy Group vs Plasma Injection Group; Test type: Superiority; p > .99, Fisher Exact

ADVERSE EVENTS:
Time Frame: Two data collection points, the second of which is between 14 and 23 days following treatment
Arm/Group | Tenotomy Group | Plasma Injection Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenotomy Group (N=15) | Plasma Injection Group (N=15)
Fever (Infections and infestations) | 0 | 1 — clinical examination showed no evidence for infection at the hip; hypothesized incidental viral origin

LIMITATIONS AND CAVEATS:
Two limitations include the small sample size and the retrospective nature of the long term secondary patient outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes